CLINICAL TRIAL: NCT00920569
Title: Measurement of Recirculation, Oxygenator Blood Volume and Cardiac Output in ECMO Using a Modified Transonic Systems (tm) HD02 Monitoring System
Brief Title: Recirculation, Oxygenator Blood Volume and Cardiac Output Measurements During Extracorporeal Membrane Oxygenation
Status: Terminated | Type: Observational
Why Stopped: Study site collaborators withdrew from participating due to time constraints.
Sponsor: Transonic Systems Inc. (Industry)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: TSI-G-HCE101-2A-H; 1R43HL082022-01 (NIH)
Record Dates: First submitted 2009-06-11; First posted 2009-06-15 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-05

CONDITIONS: Recirculation; Oxygenator Blood Volume; Cardiac Output; Venoarterial Extracorporeal Membrane Oxygenation; Venovenous Extracorporeal Membrane Oxygenation
Keywords: cardiac output; recirculation; oxygenator blood volume; venoarterial extracorporeal membrane oxygenation; venovenous extracorporeal membrane oxygenation

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is to test the usefulness of ultrasound dilution measurements in patients on extracorporeal membrane oxygenation. Measurements may include; efficiency of support (recirculation), amount of clotting in the oxygenator (oxygenator blood volume), and how well the heart is working (cardiac output). At the present time there are no devices available to perform these functions.

DETAILED DESCRIPTION:
At the present time there are no devices available to measure recirculation, oxygenator blood volume and cardiac output in patients on extracorporeal membrane oxygenation. The study uses an external monitor, laptop computer, clamp on flowsensors and ultrasound dilution technology to measure blood flow. Measurements are made by injecting 0.5 - 1 ml/kg of sterile isotonic saline into the patient's extracorporeal circuit. The subject will be monitored throughout the measurements. The measurements will be coordinated with the regular care of the extracorporeal circuit.

ELIGIBILITY:
Inclusion Criteria:

* Neonatal, pediatric or adult patients receiving venoarterial or venovenous extracorporeal membrane oxygenation.

Exclusion Criteria:

* Patients not receiving venoarterial or venovenous extracorporeal membrane oxygenation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Measurement of cardiac output in venoarterial extracorporeal membrane oxygenation patients, recirculation in venovenous extracorporeal membrane oxygenation patients and oxygenator blood volume in venoarterial and venovenous extracorporeal membrane oxygenation patients.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2006-05; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Cardiac output, recirculation or oxygenator blood volume measurements made in patients receiving extracorporeal membrane oxygenation. | Duration of extracorporeal membrane oxygenation

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Haft, MD, Principal Investigator — University of Michigan; Nikolai M Krivitski, PhD, DSc, Principal Investigator — Transonic Systems Inc.
Locations (1):
- University of Michigan, Medical School, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No